CLINICAL TRIAL: NCT02100995
Title: A Randomized Clinical Trial of an Integrated Behavioral Self-management Intervention Simultaneously Targeting Obesity and Pain: The STOP Trial
Brief Title: Simultaneously Targeting Obesity and Pain: The STOP Trial
Acronym: STOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Sciences in Philadelphia (Other)
Responsible Party: Principal Investigator, Elizabeth Amy Janke, Assistant Professor of Psychology, University of the Sciences in Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP# 4100057688
Record Dates: First submitted 2014-03-24; First posted 2014-04-01 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Obesity; Chronic Pain
MeSH Terms: conditions — Obesity; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- STOP Intervention (Experimental): The STOP treatment includes content designed to simultaneously and explicitly target both chronic pain and obesity. Treatment components are drawn from evidence-based interventions for chronic pain and obesity, separately.
  Interventions: Behavioral: Intervention Simultaneously Targeting Obesity and Pain
- Standard Care Weight (SCW) (Active Comparator): The weight loss intervention includes content focused around nutrition and eating habits, stimulus control and behavioral change, and physical activity. This content has been chosen because of its demonstrated effectiveness and importance in behavioral interventions to reduce weight.
  Interventions: Behavioral: Weight Loss/Weight Self-Management
- Standard Care Pain (SCP) (Active Comparator): The chronic pain intervention is focused around reconceptualization of pain, decreasing catastrophizing, and increasing self-efficacy for pain. This content has been chosen because of its demonstrated effectiveness and importance in non-pharmacological interventions to improve pain management.
  Interventions: Behavioral: Chronic Pain Self-Management

INTERVENTIONS:
Behavioral: Intervention Simultaneously Targeting Obesity and Pain
  Arms: STOP Intervention
Behavioral: Weight Loss/Weight Self-Management
  Arms: Standard Care Weight (SCW)
Behavioral: Chronic Pain Self-Management
  Arms: Standard Care Pain (SCP)

SUMMARY:
The purpose of this study is to determine whether an integrated behavioral treatment approach can help overweight or obese individuals who also have chronic pain reduce their weight and manage their pain symptoms. The goal of this research is to develop better treatments for individuals with chronic pain and overweight or obesity. All participants in this study will receive treatment for weight management and/or pain symptoms. Participants will be assigned at random (like we picked it blindly out of a hat) to receive either: (1) Standard behavioral treatment for weight loss; or (2) Standard behavioral treatment for pain management; or (3) Integrated behavioral treatment for weight loss and pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18
* Body mass index (BMI) ≥ 25
* Chronic, non-cancer pain (pain at a level ≥ 4 on a scale of 0-10 on a majority of the days for 6 months or more prior to study participation)

Exclusion Criteria:

* Have an unstable medical or psychiatric condition
* Meet criteria for current substance abuse or dependence
* Meet the criteria for bulimia
* Non-fluent in spoken or written English
* Currently pregnant, pregnant within the past 6 months, trying to get pregnant in the next 3 months
* Demonstrate significant cognitive or sensorimotor impairment precluding treatment engagement
* Already participating in a similar structured diet or exercise program or pain self-management program or plans to begin such a program outside the study during the next month
* At risk for significant adverse cardiovascular events with moderate activity
* Plans to relocate within the upcoming 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight from baseline to 12-months | Baseline, up to 12 months
  Body weight measured using a calibrated digital scale during assessment visits.
Change in pain intensity from baseline to 12 months | Baseline, up to 12 months
  Pain intensity as measured on a numeric ratings scale (NRS) of 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Change in pain disability from baseline to 12 months | Baseline, up to 12 months
  As measured by West Haven Yale Multidimensional Pain Inventory (WHYMPI).
Change in quality of life from baseline to 12 months | Baseline, up to 12 months
  As measured by the SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Janke, PhD, Principal Investigator — University of the Sciences in Philadelphia
Locations (1):
- University of the Sciences, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Janke EA, Fritz M, Hopkins C, Haltzman B, Sautter JM, Ramirez ML. A randomized clinical trial of an integrated behavioral self-management intervention Simultaneously Targeting Obesity and Pain: the STOP trial. BMC Public Health. 2014 Jun 18;14:621. doi: 10.1186/1471-2458-14-621. PMID 24943851